## INFORMED CONSENT FORM

## LIPID - LOWERING REGIMES IMPROVE OXIDATIVE STRESS, TRYPTOPHAN DEGRADATION IN HYPERCHOLESTEROLEMIA CKD PATIENTS

| Date of rev | view: 03 <sup>th</sup> | Mav. | 2018 |
|-------------|------------------------|------|------|
|-------------|------------------------|------|------|

| This is a research on health care, carried out by Doctor, 1 | from |
|---|---|
| Hue University of Medicine and Pharmacy. I understand that this research has been | en |
| approved by Ethnic Committee of Hue University of Medicine and Pharmacy. Su | bjects |
| of the research is: "Lipid - lowering regimes improve oxidative stress, Tryptophar | 1 |
| degradation in hypercholesterolemia CKD patients" | |

The researcher should have the patient read this form carefully and answer any questions the patient may have. Before the research can start, the researcher and the patient should sign two copies of this form. The patient will be given one copy of the signed form.

- 2. I will be randomly prescribed lipid-lowering therapy by the researcher in 12 months. I understand that there may be some side effects related to drugs such as muscle pain, muscle weakness, elevate hepatic enzyme,...My blood samples will be taken during the research, at baseline and 4, 8, 12 months of treatment.
- 3. I have to visit the clinic monthly for treatment and side effects monitoring.
- 4. My personal information and the research results related to me will be kept in secrete, not to be sent to my office and family without my permission.

| | questions or problems involved in research. |
|---|---|
| 6. | I have read and understand the explanation provided to me. I have had all my questions answered to my satisfaction, and I voluntarily agree to participate in this study. |
| For fu | orther information, please contact: Doctor |
| Date . | |
| My Signature | |
| Resea | archer Signature |